CLINICAL TRIAL: NCT06410716
Title: A Randomized Controlled Study Comparing Valve-regulated Pleural Drainage System to Traditional Closed Chest Tube Drainage
Brief Title: Comparing Valve-regulated Pleural Drainage to Traditional Closed Chest Tube Drainage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Ningbo Xinyue Medical Technology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: TDRWR-1
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: lung cancer; thoracic drainage system
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Random number table
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valve-regulated pleural drainage system (Experimental): Patients using valve-regulated pleural drainage system.
  Interventions: Device: Valve-regulated pleural drainage system
- Closed chest tube drainage (No Intervention): Patients using traditional closed chest tube drainage

INTERVENTIONS:
Device: Valve-regulated pleural drainage system — Patients using valve-regulated pleural drainage system (Ningbo Xinyue Medical Technology Co., Ltd., model AFG31-1) postoperatively.
  Arms: Valve-regulated pleural drainage system

SUMMARY:
Thoracic drainage is an important adjunctive treatment following thoracic surgery, primarily aimed at removing postoperative blood, air, and exudate from the thoracic cavity. It helps maintain negative pressure in the thoracic cavity, promotes full lung expansion, and prevents pulmonary complications, especially atelectasis. Traditional closed thoracic drainage methods have many limitations. Dry valve-regulated pleural drainage system overcome these limitations. Preliminary studies have shown that they offer advantages such as high safety, ease of operation, and reduced nursing burden. The investigators plan to conduct a real-world randomized controlled study comparing the clinical efficacy of dry valve-regulated pleural drainage system with traditional water-sealed drainage systems, both of which are commonly used in clinical practice. The goal of this study is to provide solid evidence based on evidence-based medicine for the optimal practice of thoracic drainage, further optimize post-thoracic surgery drainage treatment protocols, enhance the quality and efficiency of patient care, and provide scientific evidence for the development or updating of relevant clinical guidelines.

DETAILED DESCRIPTION:
Thoracic drainage is an important adjunctive treatment following thoracic surgery, primarily aimed at removing postoperative blood, air, and exudate from the thoracic cavity. It helps maintain negative pressure in the thoracic cavity, promotes full lung expansion, and prevents pulmonary complications, especially atelectasis. In traditional closed thoracic drainage methods, a closed drainage bottle is connected by a water-sealed tube, utilizing the pressure gradient formed by the gas-liquid interface to achieve drainage. The entire process demands high requirements for medical staff, requiring regular checks for abnormal drainage fluid, observing pressure fluctuations, and adjusting the position of the drainage bottle. This process is not only cumbersome but also carries risks of infection, drainage obstruction, and water seal fluid backflow due to operational errors.

To overcome the limitations of traditional closed drainage methods, dry valve-regulated pleural drainage systems have emerged. These devices employ a one-way valve mechanism, eliminating the need for traditional water seals and fundamentally eliminating the need for water level monitoring and maintenance of drainage bottles, while reducing the potential for mechanical failures and operational errors. They exhibit significant advantages in enhancing safety, simplifying operational procedures, and reducing nursing burdens. Patients can move more freely without worrying about water seal leakage, which is crucial for early postoperative recovery.

Preliminary prospective small-sample studies have found that compared to traditional water-sealed drainage systems, dry valve-regulated drainage devices not only significantly shorten drainage time but also reduce the need for medical staff monitoring and operation, while lowering the risk of patient pulmonary air leakage and postoperative pneumothorax. However, existing evidence mainly comes from limited hospitals and small-sample studies, lacking large-scale research to support their widespread clinical application.

Based on this, the investigators plan to conduct a real-world randomized controlled study. The study will include patients undergoing lobectomy and lymph node dissection, and different drainage methods will be randomly assigned for research. The study will compare the effects of the two thoracic drainage methods on key clinical indicators such as postoperative drainage time, drainage volume, oxyhemoglobin saturation, early postoperative activity, patient comfort during recovery, and postoperative complications. Through scientific research design and statistical analysis, the goal of this study is to provide solid evidence based on evidence-based medicine for the optimal practice of thoracic drainage, further optimize post-thoracic surgery drainage treatment protocols, and enhance the quality and efficiency of patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who accepted thoracoscopic lobectomy and lymph node dissection;
2. Written consent is able to obtained.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with significant dysfunction of organs such as the heart, liver, or kidneys;
3. Patients with pleural effusion or pneumothorax preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative drainage duration | From surgery to chest tube removal
  Postoperative drainage duration

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) cores | From surgery to chest tube removal
  The Numeric Rating Scale (NRS) will be used in assessing pain intensity of patients. The pain intensity of patients is measured on a scale from 0 to 10, with 0 representing "no pain" and 10 representing "the most intense pain".
Postoperative oxyhemoglobin saturation (SpO2) | From surgery to chest tube removal
  Postoperative drainage duration

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The research results have not been published.